CLINICAL TRIAL: NCT04330053
Title: A Record of Falls in Seniors in Central Macedonia and an Intervention for Injury Prevention Through Special Exercise Programs for Fall Prevention
Brief Title: Documentation of Fall Incidents and Application of a Fall Prevention Programme for Seniors in Northern Greece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, LYTRAS DIMITRIOS, Dimitrios Lytras PT, Phd, Postdoc Research Fellow, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44338/2020
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Elderly; Accidental Falls; Prevention; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: An assessor-blind randomized control trial with a duration of six months and a 6-month follow up will be performed in 150 seniors with a history of a previous fall. The participants will be allocated into two groups of 75 persons each (one intervention group and one control group). The first group will receive consulting about home modification for home safety related to fall prevention and training on how to avoid a fall and how to act if a fall occurs. Additionally, the first group participants will follow a fall prevention exercise program based on the OTAGO exercise program. The second group (control group) will receive only the consulting and training part excluding the fall prevention exercise program.
Who Masked: Outcomes Assessor
Masking Description: Assessor-blind randomized control trial. A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Information - Education about falls and Exercise for Fall Prevention
  Interventions: Other: Experimental
- Control (Active Comparator): Information - Education about falls without Exercise for Fall Prevention
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — * Training will address issues such as: environmental security, identifying hazards that can lead to a fall, psychological support, getting up from a fall, standing techniques and calling for help.
  * The exercise program will last for six months and will be based on the OTAGO exercise program, which includes five exercise groups: general warm-up, muscle strengthening exercises, balance exercises, range of motion and stretching exercises. The program will be performed individually or in groups of two people at most and will be conducted once a week in one of the 5 outpatient clinics under the supervision of a specialized OTAGO trainer, while seniors should repeat the exercises twice a week alone at home and also walk twice a week for at least half an hour.
  Arms: Experimental
Other: Control — * Information / Education about falls The participants in this group will receive the same information - education as the participants of the 1st group.
  * They will be given a leaflet with general gentle exercises (not fall prevention specific) for the home.
  Arms: Control

SUMMARY:
Due to the aging of the earth's population in the coming years, strategies for preventing falls in the elderly are of increasing research interest. Injuries due to falls have a direct impact on the quality of life of the elderly and are associated with very high costs for the healthcare system. However, few organized fall prevention interventions have been implemented in Greece, unlike other EU countries. The systematic recording of falls, the information and education of older people about injury prevention and the participation of older people in organized fall coping strategies in Greece are almost non-existent. Group exercise programs have proven to be effective in reducing falls. The OTAGO exercise program has shown that it can effectively reduce the number of falls in the elderly by up to 54%. However, its widespread implementation by a government agency in Greece such as the Elderly Day Care Centers (EDCC) has not yet been possible.

DETAILED DESCRIPTION:
Background: Falls in the elderly are a global health problem as they are associated with serious injuries and chronic disability. About 30% of seniors over 65 experience one or more falls each year. Any fall can lead to injury, a long period of immobilization, a decline in the functional level of the elderly, a negative psychological impact and often the elderly can even end up in death. The causes of the falls are multifactorial and are related both to the effects of aging on the human body and to environmental factors. Due to the aging of the earth's population in the coming years, strategies for preventing falls in the elderly are of increasing research interest. Injuries due to falls have a direct impact on the quality of life of the elderly and are associated with very high costs for the healthcare system. However, few organized fall prevention interventions have been implemented in Greece in contrast to other EU countries. The systematic recording of falls, the information and education of older people about injury prevention and the participation of older people in organized fall coping strategies in Greece are almost non-existent. Group exercise programs have proven to be effective in reducing falls. The combination of balance exercises and strengthening of the core and lower limbs seems to have a positive effect on the elderly in avoiding falls. The OTAGO exercise program has shown that it can effectively reduce the number of falls in the elderly by up to 54%. However, its widespread implementation by a state body has not yet been possible.

Aim: The purpose of this study is to record the incidence of falls in older people, to inform and educate them on prevention and to study the effect of specialized therapeutic exercise in relation to the usual physiotherapeutic care in reducing the number of falls. Senior people will be selected from the Elderly Day Care Centers for this purpose.

Methods / Design: About 150 elderly people over 65 are expected to participate in this study. Participants will be recruited from 15 Day Care Centers, which will be divided into two groups (intervention and control). All participants will be informed and trained in fall prevention through lectures at the Day Care Center, as well as through the distribution of appropriate audiovisual material. Subsequently, the participants of the intervention group will follow a 6-month OTAGO group exercise program, where seniors will perform exercises three times a week. The control group participants will receive a leaftlet with general exercise (not falls prevention specific). The history of falls, fear of falling, balance and functional ability of participants will be assessed before, during and after the intervention, and will be re-examined 6 months after the intervention.

Expected results: The results of this research will give a first glimpse of the magnitude of the problem of falls in older people in Greece, as data will be collected on the number of episodes, the factors that cause them, the outcome of falls, etc. The effectiveness of targeted exercise programs and in particular of OTAGO in reducing the number of falls and improving the balance and functional capacity of older people will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 - 80
* Ambulatory people who walk independently or with some walking assistance device
* People with a history of at least one fall in the last 12 months
* People with Timed Up and Go test score minor than 15sec

Exclusion Criteria:

* People who were diagnosed with neurodegenerative disease (e.g. Parkinson's disease)
* People who recently had a stroke
* People with decreased ability to communicate (senile dementia etc.)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Changes in CONFbal - GREEK score questionnaire | Pre-treatment, Month 6, 12
  The CONFbal questionnaire is a tool that assesses the self-esteem of an elderly person associated with the risk of falling. It consists of a 10-item scale, which are summed to give an index of balance confidence. The score ranges from 10 to 30. A higher score indicates lower balance confidence. Τhe questionnaire demonstrates excellent internal consistency and excellent test-retest reliability. The Greek version of the questionnaire CONFbal - GREEK (Billis, et al., 2011) will be used in this study.
Changes in Short Falls Efficacy Scale International (Short FES-I) score questionnaire | Pre-treatment, Month 6, 12
  Short FES-I is a measure of "fear of falling" or, more properly, "concerns about falling", which are suitable for use in research and clinical practice. It is the short version of the Falls Efficacy Scale International (FES-I), comprised of seven questions and is more applicable in clinical practice. The score ranges from 7 to 28. A higher score indicates greater fear of falling. The Greek version of the questioner (Billis, et al., 2011) will be used in this study
Changes in 4-Stage Balance Scale test | Pre-treatment, Month 6, 12
  The 4-Stage Balance Test is an assessment of static balance in four different and increasingly challenging positions - feet together, instep of foot advanced to toe of other foot, foot in front of other foot (tandem), and single leg stance (Lajoie & Gallagher, 2004). The participant must stand in each position for ten seconds, while the examiner tracks time using a stopwatch. Each of the first three positions is evaluated with the eyes open and closed, while the single leg stance is evaluated only with the eyes open, so each participant is evaluated in a total of seven tests. Each test is scored from four to zero (representing "able to stand for 10 seconds safely" and "needs help to keep from falling" respectively). The final score results from the sum of all seven tests and ranges from zero to 28. A higher score indicates greater static balance ability of the participant. The test has good validity (Marques et al., 2017).
Changes in Timed Up and Go test | Pre-treatment, Month 6, 12
  It is a simple test used to assess a person's mobility. It requires both static and dynamic balance and is a valid and reliable indicator of the functional ability of an individual (Podsiadlo & Richardson). The participant starts in a seated position. They then stand up following the instructions of the therapist, walk three meters, turn around, walk back to the chair and sit down. The examiner tracks time using a stopwatch. Time is calculated in seconds. A higher score indicates lower functional ability of the participant.
Changes in number of falls | Pre-treatment, Month 6, 12
  Changes in number of falls will be evaluated through a Falls diary which will be completed each month by the elderly
Changes in the 30-Second Chair Stand Test | Pre-treatment, Month 6, 12
  The 30-Second Chair Stand Test is a test for assessing leg strength and endurance in elderly adults. It is part of the Stop Elderly Accidents, Deaths, and Injuries (STEADI) tool kit, which was created by the Centers for Disease Control and Prevention as a screening tool for seniors belonging in the high fall risk group (Stevens, 2013). The test measures the number of times an elderly person can get up from a chair with their arms crossed in front of their trunk (on the opposite shoulder crossed at the wrists) in 30sec. This test was developed to overcome the floor effect of the five or ten repetition sit to stand test in older adults. The test has been characterized by excellent test-retest reliability in a total number of participants: r = 0.89 (95% Confidence interval 0.79-0.93) (Rikli & Jones, 1999).
Changes in Berg Balance scale Test | Pre-treatment, Month 6, 12
  The Berg Balance Scale is a tool proposed by Berg (Berg et al., 1989; Berg et al., 1992) for assessing balance in the elderly. The test involves the execution of 14 tests of gradual increasing difficulty where in each one, the subject is asked to maintain a given position for a specific time or conduct specific tasks. Each of the 14 tests on the list is graded according to the balancing ability of the examinee from 0 to 4 points (with 0 indicating low balance ability, while 4 indicates high balance ability). According to Berg et al. (1992), a score of 56 indicates functional balance, whereas a score lower than 45 indicates notable balance deficits that have been related to increased fall risk. Studies have shown high intra-rater and inter-rater reliability in the elderly populations with intraclass correlation (ICC) ranging from .98 to .88 (Berg et al. 1992) and high content validity (Telenius et al., 2015).

SECONDARY OUTCOMES:
Changes in adherence to exercise via Exercise Diary keeping | Month 7, 8, 9, 10, 11, 12
  After the 6 months intervention period the participants of both groups will be asked to continue to perform the specific exercise programs three times per week for a period of six months recording the adherence or not to the exercise programs in a weekly diary while the assessor will collect the data by phone 2-3 times a month.

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Sykaras, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Central Makedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lytras D, Sykaras E, Iakovidis P, Komisopoulos C, Chasapis G, Mouratidou C. Effects of a modified Otago exercise program delivered through outpatient physical therapy to community-dwelling older adult fallers in Greece during the COVID-19 pandemic: a controlled, randomized, multicenter trial. Eur Geriatr Med. 2022 Aug;13(4):893-906. doi: 10.1007/s41999-022-00656-y. Epub 2022 May 24. PMID 35606677